CLINICAL TRIAL: NCT05256394
Title: Scaling Interoperable Clinical Decision Support for Patient-Centered Chronic Pain Care
Brief Title: Patient-Centered Chronic Pain Care
Acronym: IPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB202101931; 1R18HS028584-01 (AHRQ)
Record Dates: First submitted 2022-01-28; First posted 2022-02-25 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pain; Opioid Use; Musculoskeletal Pain
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: This is a stepped-wedge, cluster randomized trial using mixed methods to assess the multilevel determinants of CDS implementation success. The investigators will use both quantitative and qualitative data to provide a comprehensive understanding of the clinical context of the participating sites before and after the trial, and identify system, clinic and provider-level factors that may influence the implementation process. In summary, this is a complete, open-cohort stepped-wedge cluster-randomized design with 5 time periods (including the baseline), with each period spanning 1 month and 2 clinics switching from control to intervention at each of the 4 steps (for a total study duration of 5 months).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Manager + tailored implementation support Pain Manager (Active Comparator): Pain Manager is a decision support tool. All study clinics will begin the trial with Pain Manager integrated and available in their EHR. Consistent with the stepped-wedge design, intensive implementation support (e.g, administrative support, technical support)will be provided to two clinics at once by a multidisciplinary team.
  Interventions: Behavioral: Pain Manager + tailored implementation support
- Pain Manager implementation in EHR (No Intervention): Pain Manager is a decision support tool. All study clinics will begin the trial with Pain Manager integrated and available in their EHR. The other 6 clinics will have no additional tailor support.

INTERVENTIONS:
Behavioral: Pain Manager + tailored implementation support — Individualized training, technical assistance, and workflow assessments.
  Arms: Pain Manager + tailored implementation support Pain Manager

SUMMARY:
This study will adapt and scale existing AHRQ-supported interoperable CDS for patient-centered chronic pain care. The objective of this project is to study the adaptation and implementation of an existing interoperable CDS tool for pain treatment shared decision making, with tailored implementation support, in primary care clinical settings. The central hypothesis is that tailored implementation support will increase CDS adoption and shared decision making.

DETAILED DESCRIPTION:
This study will adapt and scale the use of existing AHRQ-supported interoperable CDS that aids patient-centered chronic pain treatment decision making. The research will generate critical evidence on scalable strategies to implement and evaluate interoperable CDS in real-world settings across different types of EHRs. The pragmatic trial will enhance the reach of interoperable CDS to more diverse populations. Together, these efforts will lead to important new technology and evidence that patients, clinicians, and health systems can use to improve care for millions of Americans who suffer from pain and other chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Primary care patients receiving care at a participating clinic
* Patients with chronic non-cancer musculoskeletal pain and with a recent history of opioid use

Exclusion Criteria:

* Due to the fact that the clinical decision support tool is currently available in English only, non-English speaking patients will not be eligible to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Adoption | During the implementation trial (5 months total)
  Rate of qualifying patients seen for whom CDS use is documented

SECONDARY OUTCOMES:
Reach | During the implementation trial (5 months total)
  Rate of clinic encounters where CDS is documented
Shared decision making | Immediately after the intervention
  SDM-Q-9 questionnaire: 9-item Shared Decision Making Questionnaire
Pain and function | Baseline/pre-intervention, and at 1 and 3 months
  PEG-3: 3-item scale that measures pain on average, its interference with enjoyment of life, and with general activity
Any opioid prescription | Baseline/pre-intervention, and at 1 and 3 months
  Binary measure of treatment choice that increases opioid-related risks
Opioid prescriptions ≥50 MME/day | Baseline/pre-intervention, and at 1 and 3 months
  Binary measure of treatment choice that increases opioid-related risks
Opioid prescriptions ≥90 MME/day | Baseline/pre-intervention, and at 1 and 3 months
  Binary measure of treatment choice that increases opioid-related risks
Benzodiazepine prescription concurrent with opioid prescription | Baseline/pre-intervention, and at 1 and 3 months
  Binary measure of treatment choice that increases opioid-related risks
Prescriptions for non-opioid pain medications | Baseline/pre-intervention, and at 1 and 3 months
  Binary measure recommended by the CDC to decrease opioid-related risks
Prescriptions for non-pharmacologic pain treatments | Baseline/pre-intervention, and at 1 and 3 months
  Binary measure recommended by the CDC to decrease opioid-related risks
Urine drug screen orders | Baseline/pre-intervention, and at 1 and 3 months
  Binary measure recommended by the CDC to decrease opioid-related risks
Naloxone prescriptions | Baseline/pre-intervention, and at 1 and 3 months
  Binary measure recommended by the CDC to decrease opioid-related risks
Prescription or referral for medication-assisted therapy (MAT) | Baseline/pre-intervention, and at 1 and 3 months
  Binary measure recommended by the CDC to decrease opioid-related risks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Harle, Ph.D., Principal Investigator — University of Florida
Locations (1):
- UF Health Family Medicine - Commonwealth, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salloum RG, Bilello L, Bian J, Diiulio J, Paz LG, Gurka MJ, Gutierrez M, Hurley RW, Jones RE, Martinez-Wittinghan F, Marcial L, Masri G, McDonnell C, Militello LG, Modave F, Nguyen K, Rhodes B, Siler K, Willis D, Harle CA. Study protocol for a type III hybrid effectiveness-implementation trial to evaluate scaling interoperable clinical decision support for patient-centered chronic pain management in primary care. Implement Sci. 2022 Jul 15;17(1):44. doi: 10.1186/s13012-022-01217-4. PMID 35841043

DOCUMENTS (1):
  • Informed Consent Form (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT05256394/ICF_000.pdf